CLINICAL TRIAL: NCT02397538
Title: An Open-label, Fixed-sequence, Crossover Study to Evaluate the Pharmacokinetic Interaction and Safety After Multiple Oral Doses of Fimasartan/Amlodipine and Rosuvastatin in Healthy Male Subjects
Brief Title: Study to Evaluate the Pharmacokinetic Interaction and Safety After Multiple Oral Doses of Fimasartan/Amlodipine and Rosuvastatin in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Inje University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BR-FARC-CT-101
Record Dates: First submitted 2015-03-16; First posted 2015-03-25 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-03

CONDITIONS: Hypertension
Keywords: Fimasartan
MeSH Terms: conditions — Hypertension | interventions — fimasartan; Amlodipine; Rosuvastatin Calcium

ARMS (2):
- Cohort1 (Other): Treatment AB → ABC Treatment A+B (10days) → Treatment A+B+C (6days) Treatment A: Fimasartan Treatment B: Amlodipine Treatment C: Rosuvastatin
  Interventions: Drug: Fimasartan; Drug: Amlodipine; Drug: Rosuvastatin
- Cohort2 (Other): Treatment C → ABC Treatment C (6days) → Treatment A+B+C (10days) Treatment A: Fimasartan Treatment B: Amlodipine Treatment C: Rosuvastatin
  Interventions: Drug: Fimasartan; Drug: Amlodipine; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Fimasartan
Drug: Amlodipine
Drug: Rosuvastatin

SUMMARY:
An Open-label, Fixed-sequence, Crossover Study to Evaluate the Pharmacokinetic Interaction and Safety after multiple oral doses of Fimasartan/Amlodipine and Rosuvastatin in Healthy Male Subjects.

DETAILED DESCRIPTION:
After subjects have signed informed consent voluntarily, they go through screening period for within 28 days.

As period I, subjects of Cohort1 take fimasartan and Amlodipine for 10 days and subjects of Cohort2 take rosuvastatin for 6 days.

And then, as period II, subjects of both Cohorts take fimasartan, Amlodipine and rosuvastatin in Cohort1 case for 6 days and in Cohort2 case for 10 10days.

For Fimasartan, subjects of Cohort1 have blood sampling 8th, 9th, 14th, 15th day before medication, 10th and 16th day before and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 and 24hour after medication(32 times in total).

For Amlodipine, subjects of Cohort1 have blood sampling 8th, 9th, 14th, 15th day before medication, 10th and 16th day before and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 24hour after medication(30 times in total).

For Rosuvastatin and N-desmethyl rosuvastatin, subjects of Cohort2 have blood sampling 4th, 5th, 14th, 15th day before medication, 6th and 16th day before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12 and 24hour after medication(28 times in total).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subject, aged 19- 50 years at screening.
2. Body weight within ± 20% of ideal body weight (IBW)(kg) = {height (cm) - 100} * 0.9

Exclusion Criteria:

1. History of any illness that may affect the absorption, distribution, metabolism or excretion (hepatobiliary, renal, cardiovascular, endocrine (e.g., hypothyroidism), respiratory, gastrointestinal, hemato-oncology, central nervous system, psychiatric and musculoskeletal system)
2. Hypotension (systolic ≤ 100 mmHg or diastolic ≤ 65 mmHg) or hypertension (systolic ≥ 140 mmHg or diastolic ≥ 90 mmHg), measured at screening
3. Active liver disease, or the levels of ALT(Aspartate Transaminase), AST (Alanin Transaminase) or total bilirubin > 1.25 x the upper limit of normal
4. History of gastrointestinal disease (i.g., Crohn's disease, active peptic ulcer) or resection operation that may affect the absorption of the study drug (excluding simple appendectomy or herniorrhaphy)]
5. Participation in any other study within 3 months prior to the first administration of study drug (The finish time of previous study is the day of the last administration of study drug)

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Cmax,ss | Time Frame: 0~24 hour after medication
  When 1 cohort, it's a measure on Fimasartan and Amlodipine. and when another cohort, it's a measure on Rosuvastatin
AUC tau,ss | Time Frame: 0~24 hour after medication
  When 1 cohort, it's a measure on Fimasartan and Amlodipine. and when another cohort, it's a measure on Rosuvastatin

CONTACTS AND LOCATIONS:
Locations (1):
- Inje University Busan Paik Hospital, Busan, Korea, Republic of, South Korea